CLINICAL TRIAL: NCT00930319
Title: Effectiveness and Safety of Firmagon® in Androgen Ablative Therapy of Advanced Hormone-dependent Prostate Carcinoma
Brief Title: Effectiveness and Safety of Firmagon®
Acronym: FAST
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: FE200486 CS41
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2014-03

CONDITIONS: Androgen Ablative Therapy of Advanced Hormone-dependent Prostate Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Advanced Hormone-dependent Prostate Carcinoma treated with Firmagon according to SPC
  Interventions: Other: Firmagon given by prescription according to SPC

INTERVENTIONS:
Other: Firmagon given by prescription according to SPC — Non-interventional,observational Firmagon given by prescription according to SPC

SUMMARY:
Effectiveness and Safety of Firmagon® in Androgen Ablative Therapy of Advanced Hormone-dependent Prostate Carcinoma. The period until Prostate Specific Antigen (PSA) progression during the Firmagon® therapy is to be documented and related to the testosterone values measured in the course of therapy (if available). Other clinical parameters, the patients' quality of life and the direct and indirect costs incurred by the medical care for the advanced hormone-dependent prostate carcinoma and its consequences will be evaluated. In this context the medical outcome and the life quality are defined as effectiveness and benefit value parameters. Both the effectiveness under daily life circumstances and economic variables of the therapy can thus be shown and compared within an analysis of costs vs. benefits or costs vs. effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* therapeutic need according to SPC
* written informed consent

Exclusion Criteria:

- contraindications according to SPC

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Advanced Hormone-dependent Prostate Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
duration of the PSA progression-free survival | open (until therapy end or stop)

SECONDARY OUTCOMES:
1. testosterone levels | open (until therapy end or stop)
2. number of ADRs and SUSARs | open (until therapy end or stop)
3. quality of life | open (until therapy end or stop)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (230):
- Germany (230):
  - Investigational Site, Heinrich-Rieger-Str. 15, Aalen
  - Investigational Site, Weidenfelder Straße 1, Aalen
  - Investigational Site, Abensberg
  - Investigational Site, Ahaus
  - Investigational Site, Ahrensburg
  - Investigational Site, Alsdorf
  - Investigational Site, Alsfeld
  - Investigational Site, Altenburg
  - Investigational Site, Andernach
  - Investigational Site, Endresstraße 12, Ansbach
  - Investigational Site, Platenstraße 15, Ansbach
  - Investigational Site, Frölichstraße 13, Augsburg
  - Investigational Site, Prinzregentenstraße 4, Augsburg
  - Investigational Site, Bad Bergzaben
  - Investigational Site, Bad Godesberg
  - Investigational Site, Bad Marienberg
  - Investigational Site, Bad Oldesloe
  - Investigational Site, Bad Salzuflen
  - Investigational Site, Bad Schönborn
  - Investigational Site, Bad Wildungen
  - Investigational Site, Bautzen
  - Investigational Site, Albert-Einstein-Straße 2, Berlin
  - Investigational Site, Allee der Kosmonauten 47, Berlin
  - Investigational Site, Hohenzollerndamm 47a, Berlin
  - Investigational Site, Lipschitzallee 20, Berlin
  - Investigational Site, Mehrower Allee 22, Berlin
  - Investigational Site, Pasteurstraße 8, Berlin
  - Investigational Site, Rudolff-Seifert-Straße 11, Berlin
  - Investigational Site, Wisbyer Straße 16, Berlin
  - Investigational Site, Zeppelinring 7, Biberach
  - Investigational Site, Biedenkopf
  - Investigational Site, Elbeallee 83, Bielefeld
  - Investigational Site, Friedrich-Verleger Straße 5, Bielefeld
  - Investigational Site, Johannisstraße 43, Bielefeld
  - Investigational Site, Treppenstraße 3, Bielefeld
  - Investigational Site, Bitterfeld-Wolfen
  - Investigational Site, Bocholt
  - Investigational Site, St. Augustiner-Straße 21, Bonn
  - Investigational Site, Trierer Straße 70 - 72, Bonn
  - Investigational Site, Borken
  - Investigational Site, Bramsche
  - Investigational Site, Braunschweig
  - Investigational Site, Bremen
  - Investigational Site, Dr.-Franz-Mertens-Straße 8, Bremerhaven
  - Investigational Site, Georgstraße 44, Bremerhaven
  - Investigational Site, Bruchköbel
  - Investigational Site, Buchholz
  - Investigational Site, Burg
  - Investigational Site, Bünde
  - Investigational Site, Celle
  - Investigational Site, Carl-von-Ossietzky-Str. 151, Chemnitz
  - Investigational Site, Clausstraße 44, Chemnitz
  - Investigational Site, Flemmingstraße 1b, Chemnitz
  - Investigational Site, Unritzstraße 21 c, Chemnitz
  - Investigational Site, Coburg
  - Investigational Site, Custodistraße 3-17, Cologne
  - Investigational Site, Wilhelm-Ewald-Weg 1, Cologne
  - Investigational Site, Zeppelinstraße 1, Cologne
  - Investigational Site, Cottbus
  - Investigational Site, Karlstraße 30, Crailsheim
  - Investigational Site, Postplatz 2, Crailsheim
  - Investigational Site, Delitzsch
  - Investigational Site, Dessau
  - Investigational Site, Dillenburg
  - Investigational Site, Dinslaken
  - Investigational Site, Dortmund
  - Investigational Site, Dossenheim
  - Investigational Site, Dresden
  - Investigational Site, Kreuzstraße 3-5, Duisburg
  - Investigational Site, Königstraße 49, Duisburg
  - Investigational Site, Dülmen
  - Investigational Site, Düsseldorf
  - Investigational Site, Eisenhüttenstadt
  - Investigational Site, Geschwister-Scholl-Str. 6, Erfurt
  - Investigational Site, Juri-Gagarin-Ring 94, Erfurt
  - Investigational Site, Essen
  - Investigational Site, Finsterwalde
  - Investigational Site, Eschersheimer Landstr. 544, Frankfurt
  - Investigational Site, Im Steinbügel 13, Frankfurt
  - Investigational Site, Freiburg im Breisgau
  - Investigational Site, Freital
  - Investigational Site, Friedberg
  - Investigational Site, Friedrichshafen
  - Investigational Site, Arminstraße 24, Gelsenkirchen
  - Investigational Site, Feldmarkstraße 109, Gelsenkirchen
  - Investigational Site, Zum Ehrenmal 21, Gelsenkirchen
  - Investigational Site, Gera
  - Investigational Site, Giessen
  - Investigational Site, Helenenstraße 10-12, Gotha
  - Investigational Site, Schützenberg 10, Gotha
  - Investigational Site, Grimma
  - Investigational Site, Niemeyerstraße 23, Halle
  - Investigational Site, Reilstraße 129 a, Halle
  - Investigational Site, Steinweg 27, Halle
  - Investigational Site, Alte Holstenstraße 16, Hamburg
  - Investigational Site, Fuhlsbüttler Straße 182, Hamburg
  - Investigational Site, Grindelberg 3, Hamburg
  - Investigational Site, Herthastraße 12, Hamburg
  - Investigational Site, Tangstedter Landstraße 77, Hamburg
  - Investigational Site, Hattersheim
  - Investigational Site, Heidelberg
  - Investigational Site, Heilbronn
  - Investigational Site, Heinsberg
  - Investigational Site, Hennigsdorf
  - Investigational Site, Herford
  - Investigational Site, Enoch-Widmann-Straße 5, Hof
  - Investigational Site, Eppenreuther Straße 28, Hof
  - Investigational Site, Isenburg
  - Investigational Site, Jena
  - Investigational Site, Jülich
  - Investigational Site, Kaiserslautern
  - Investigational Site, Kamenz
  - Investigational Site, Kamp-Lintfort
  - Investigational Site, Karlsruhe
  - Investigational Site, Kempten
  - Investigational Site, Markt 11, Kiel
  - Investigational Site, Prüner Gang 15, Kiel
  - Investigational Site, Schulstraße 7, Kiel
  - Investigational Site, Kleinblittersdorf
  - Investigational Site, Friederikenstraße 30, Köthen
  - Investigational Site, Siebenbrünnenpromenade 6-7, Köthen
  - Investigational Site, Krefeld
  - Investigational Site, Kulmbach
  - Investigational Site, Lampertheim
  - Investigational Site, Langenau
  - Investigational Site, Lebach
  - Investigational Site, Leutkirch
  - Investigational Site, Lichtenfels
  - Investigational Site, Limbach-Oberfrohna
  - Investigational Site, Lubnjow
  - Investigational Site, Ludwigshafen
  - Investigational Site, Lübeck
  - Investigational Site, Lüneburg
  - Investigational Site, Lünen
  - Investigational Site, Magdeburg
  - Investigational Site, Mainz
  - Investigational Site, N7, 9, Mannheim
  - Investigational Site, Seckenheimer Hauptstraße 107, Mannheim
  - Investigational Site, Marburg
  - Investigational Site, Marl
  - Investigational Site, Mechernich
  - Investigational Site, Merseburg
  - Investigational Site, Merzig
  - Investigational Site, Michelstadt
  - Investigational Site, Miltenberg
  - Investigational Site, Moers
  - Investigational Site, Mölln
  - Investigational Site, Mörlenbach
  - Investigational Site, Mühlacker
  - Investigational Site, Mühlhausen
  - Investigational Site, Mühlheim
  - Investigational Site, Fürstenbergstraße 5, Münster
  - Investigational Site, Hohenzollernring 70, Münster
  - Investigational Site, Naumburg
  - Investigational Site, Neu-Ulm
  - Investigational Site, Neunkirchen
  - Investigational Site, Neuss
  - Investigational Site, Nienburg
  - Investigational Site, Norderstedt
  - Investigational Site, Bahnhofstraße 17, Nordhausen
  - Investigational Site, Bahnhofstraße 8, Nordhausen
  - Investigational Site, Am Museumsturm 4, Nordhorn
  - Investigational Site, Osnabrücker Straße 1, Nordhorn
  - Investigational Site, Am Stadtpark 2, Nuremberg
  - Investigational Site, Hefnersplatz 1, Nuremberg
  - Investigational Site, Kopernikusplatz 7, Nuremberg
  - Investigational Site, Obernburg
  - Investigational Site, Ochsenfurt
  - Investigational Site, Offenbach
  - Investigational Site, Osnabrück
  - Investigational Site, Paderborn
  - Investigational Site, Pasewalk
  - Investigational Site, Pirna-Copitz
  - Investigational Site, Prüm
  - Investigational Site, Pulheim
  - Investigational Site, Hindenburgstraße 10 A, Rastatt
  - Investigational Site, Kaiserstraße 7, Rastatt
  - Investigational Site, Gartenstraße 22, Ravensburg
  - Investigational Site, Grüner-Turm-Straße 7-9, Ravensburg
  - Investigational Site, Regensburg
  - Investigational Site, Remscheid
  - Investigational Site, Ribnitz-Damgarten
  - Investigational Site, Große Wasserstraße 2 - 3, Rostock
  - Investigational Site, Nobelstraße 51, Rostock
  - Investigational Site, Trelleborger Straße 10B, Rostock
  - Investigational Site, Rottweil
  - Investigational Site, Röthenbach an der Pegnitz
  - Investigational Site, Mainzer Straße 105, Saarbrücken
  - Investigational Site, Viktoriastraße 2, Saarbrücken
  - Investigational Site, Saarlouis
  - Investigational Site, Salzmünde
  - Investigational Site, Schönebeck
  - Investigational Site, Schwandorf in Bayern
  - Investigational Site, Schwäbisch Gmünd
  - Investigational Site, Schwerin
  - Investigational Site, Schwerte
  - Investigational Site, Senden
  - Investigational Site, Sindelfingen
  - Investigational Site, Sömmerda
  - Investigational Site, Kirchplatz 6a, Spremberg
  - Investigational Site, Lustgartenstraße 3, Spremberg
  - Investigational Site, Stockelsdorf
  - Investigational Site, Stolberg
  - Investigational Site, Stuttgart
  - Investigational Site, Sulzbach-Rosenberg
  - Investigational Site, Tettnang
  - Investigational Site, Tostedt
  - Investigational Site, Trier
  - Investigational Site, Troisdorf
  - Investigational Site, Hirschstraße 22, Ulm
  - Investigational Site, Olgastraße 103, Ulm
  - Investigational Site, Olgastraße 139, Ulm
  - Investigational Site, Überlingen
  - Investigational Site, Velbert
  - Investigational Site, Völklingen
  - Investigational Site, VS-Villingen
  - Investigational Site, Wangen
  - Investigational Site, Moosbürger Str. 13, Weiden
  - Investigational Site, Postgasse 1, Weiden
  - Investigational Site, Weißenfels
  - Investigational Site, Werl
  - Investigational Site, Werningerode
  - Investigational Site, Wesel
  - Investigational Site, Wiesbaden
  - Investigational Site, Wilhelmshaven
  - Investigational Site, Heinrich-Nordhoff-Straße 49, Wolfsburg
  - Investigational Site, Porschestraße 100, Wolfsburg
  - Investigational Site, Würselen
  - Investigational Site, Xanten
  - Investigational Site, Zerbst